CLINICAL TRIAL: NCT07275541
Title: Platelet Aggregation in the Diagnosis of Acute Graft Rejection
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Martin (Other)
Responsible Party: Principal Investigator, Matej Vnucak, ass. prof., Deputy Head of Transplant-Nephrology Department, University Hospital, Martin
Other Study IDs: TNO_AGRE; UK/3248/2024 (Other Grant/Funding Number: CU Grant - EXCELLENT 2024)
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Platelet Aggregation; Kidney Transplant Rejection
Keywords: kidney transplantation; platelet aggregation; acute rejection; non-invasive marker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- kidney transplant recipients - Protocol Biopsy Cohort: Adult kidney transplant recipients undergoing routine protocol biopsies at 3 and 12 months post-transplant, regardless of clinical graft function. Platelet aggregation, flow-cytometric P-selectin expression, soluble P-selectin levels, and biochemical and immunological parameters are collected at each time point.
  Findings from platelet function testing are subsequently correlated with the histopathological results of the protocol biopsy, including the presence or absence of subclinical rejection.
- kidney transplant recipients - Indication Biopsy Cohort: Kidney transplant recipients presenting with clinical signs of graft dysfunction-such as rising serum creatinine, increasing proteinuria, or abnormal ultrasound findings or with newly positive donor-specific antibodies (DSA) detected by Luminex testing, prompting the need for an indication biopsy due to suspected acute rejection. At the time of biopsy, platelet aggregation testing, P-selectin markers, comprehensive biochemical parameters, and DSA levels are collected. This cohort represents patients with clinically or immunologically apparent graft injury, allowing comparison with protocol-biopsied patients, including those with subclinical or biopsy-confirmed rejection.

SUMMARY:
The study titled "Platelet Aggregation in the Diagnosis of Acute Graft Rejection" is a pilot observational study evaluating whether alterations in platelet function can serve as non-invasive markers of acute rejection in kidney transplant recipients. Platelet aggregation is assessed using optical aggregometry, flow-cytometric P-selectin (CD62-P) expression, and soluble P-selectin levels before kidney transplantation and at the time of protocol biopsies performed at 3 and 12 months after kidney transplantation. Patients with suspected graft dysfunction undergoing indication biopsy are also included. Platelet activation markers are correlated with histopathological findings, donor-specific antibodies, metabolic parameters, and clinical outcomes. The goal is to determine whether platelet activation profiles can identify acute cellular or antibody-mediated rejection and contribute to the development of a non-invasive diagnostic tool.

DETAILED DESCRIPTION:
Platelets play a key role not only in hemostasis but also in inflammation and immune responses. Their activation, characterized by adhesion, integrin-mediated aggregation, thromboxane A₂ production, and surface expression of markers such as P-selectin, contributes to interactions with T lymphocytes and amplification of immune signaling. Emerging evidence suggests that platelet activation may participate in early mechanisms of kidney graft injury. Studies have demonstrated platelet accumulation in glomerular and peritubular capillaries during antibody-mediated rejection, likely mediated by donor-specific antibodies and endothelial activation via von Willebrand factor. Elevated platelet activation markers such as PF4 and P-selectin have also been associated with T-cell-mediated rejection.

This pilot study investigates whether changes in platelet aggregation and platelet activation markers can serve as non-invasive indicators of acute kidney allograft rejection. Platelet function is measured using optical aggregometry, flow cytometry of P-selectin (CD62-P), and soluble P-selectin levels. These parameters are correlated with histological findings from protocol biopsies at 3 and 12 months post-transplant, as well as from indication biopsies performed for suspected rejection. The study includes adult kidney transplant recipients monitored longitudinally and a cohort of patients with graft dysfunction requiring indication biopsy. Concurrent assessments include renal function, donor-specific antibodies, levels of immunosupression (tacrolimus), metabolic parameters, and imaging. By comparing platelet activation profiles with biopsy-proven rejection, the study aims to determine whether platelet-based biomarkers can support early, non-invasive detection of cellular or antibody-mediated allograft injury and complement traditional biopsy-based diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years)
* primary kidney transplantation
* living / deceased donor kidney transplantation
* ability and consent to participate

Exclusion Criteria:

* non-adult patients
* secondary / tertiary kidney transplantation
* antiplatelet therapy
* patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease who underwent kidney transplantation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-11-26 (Estimated); Study Completion 2027-11-26 (Estimated)

PRIMARY OUTCOMES:
To compare changes in platelet aggregation in patients before and after kidney transplantation | Pre-transplant baseline; 3 months post-transplant; 12 months post-transplant
  Platelet aggregation measured by optical aggregometry before kidney transplantation will be compared with platelet aggregation measured at 3 and 12 months after transplantation to assess changes in platelet function over time.
To evaluate the changes in platelet aggregation in the diagnosis of humoral/cellular graft rejection (at the time of biopsy due to graft dysfunction) | At the time of indication biopsy (any time after transplantation)
  Platelet aggregation will be assessed at the time of an indication biopsy performed for graft dysfunction and compared between patients with biopsy-proven humoral or cellular rejection and those without rejection. The aim is to determine whether altered platelet aggregation is associated with acute graft rejection identified on histopathology.
To investigate the use of P-selectin as a potential marker of platelet activation in the diagnosis of acute graft rejection as part of a non-invasive investigation | Pre-transplant baseline; at 3- and 12-month protocol biopsies; and at the time of any indication biopsy after kidney transplantation
  Flow-cytometric P-selectin (CD62-P) expression on platelets and soluble P-selectin levels in plasma will be measured before and after kidney transplantation and at the time of protocol or indication biopsy. These values will be compared between patients with and without biopsy-proven rejection to assess whether P-selectin can serve as a reliable marker of platelet activation associated with acute graft injury and support the development of a non-invasive diagnostic approach.

CONTACTS AND LOCATIONS:
Overall Officials: Matej Vnucak, ass prof, MD, PhD., Study Chair — University Hospital Martin and Jessenius Faculty of Medicine, Comenius University
Locations (1):
- Transplant-Nephrology Department, University Hospital Martin, Martin, Slovakia

IPD SHARING:
Plan to Share IPD: No
It is a monocenter pilot study